CLINICAL TRIAL: NCT02046876
Title: Swimming Adapted, Therapeutic Exercise and Health Education in the Treatment of Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UMA-1301
Record Dates: First submitted 2013-12-24; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Neck Pain
Keywords: neck pain; physiotherapy; adapted swimming; therapeutic exercises; health education
MeSH Terms: conditions — Neck Pain; Health Education

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multimodal Physiotherapy Program for Chronic Neck Pain Suffers (Experimental)
  Interventions: Other: Multimodal Physiotherapy Program

INTERVENTIONS:
Other: Multimodal Physiotherapy Program — Multimodal Physiotherapy Program integrates: physical land-based therapeutic exercise, adapted swimming and health education

SUMMARY:
Chronic neck pain (CNP) is defined as pain or intense discomfort in the lateral or back of the neck with an establishment and/or persistence period of over 12 weeks.

The socio-economic system is seriously affected by chronic neck pain due to direct and indirect costs on the health system Physical exercise is used to improve physical function and reduce the symptoms of pain and stiffness due to chronic neck pain.

It has been demonstrated that therapeutic exercise in water is effective to improve functional capacity and symptoms in patients with chronic neck pain. In adition, health education and posture is an important component of the overall treatment of neck pain.

Interventions that integrate physical activity, adapted swimming and health education as an intervention for chronic neck pain sufferers have not been found. Furthermore the aim of this study is to analyse the effect of a physiothperapy treatment that combine adapted swimming, therapeutic exercise and health education in patients with chronic neck pain.

Hypothesis: the present intervention will be an effective tool to treat patients suffering chronic neck pain.

Methods: chronic neck pain patients from a community-based centre will be recruite participate in this prospective study.

Intervention: 60 min session: 30 min of land exercise dedicated to improve mobility, motor control, resistance and strengthening of the neck muscles, 30 min of adapted swimming with aerobic exercise keeping neutral neck position by using a snorkel. Health education will be provided by the physiotherapist before and during the sessions using a decalogue on chronic neck pain and constant repetition of brief advice.

Study outcomes: disability (Neck Disability Index), physical and mental health state and quality of life of patients (SF-12 and EuroQoL 5D respectively).

Differences between baseline data and that at the 8-week follow-up were calculated for all outcome variables.

Statistical Analysis: descriptive statistics. Analysis of the normal distribution of the variables using the KS-test. Comparison of variables pre - post intervencición: T-Student for parametric variables and Wilcoxon test for non parametric variables.

Data will be analysed descriptively and for statistical significance using Statistical Package for the Social Sciences (SPSS) (version 17.0 for Windows, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* Suffers Neck Pain for more than 12 weeks.
* Delivery of informed consent.

Exclusion Criteria:

* Neck pain due to an identifiable cause.
* Surgery on the spine in the 12 month
* Traffic accident in the last 3 months
* Cervical radiculopathy
* Pregnancy.
* Patients who suffered a condition that could alter the effects of treatment
* People who could not swim and/or present treatment difficulty.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Change from baseline in NDI at 8 weeks (post-treatment)
  Disability due to Chonic Neck Pain
Neck Disability Index | Change from baseline in NDI at 6 month (follow-up)
  Disability due to Chonic Neck Pain
Neck Disability Index | Change from baseline in NDI at 12 month (follow-up)
  Disability due to Chonic Neck Pain

SECONDARY OUTCOMES:
Short Form 12 | pre and post intervention and 6 and 12 months of follow up
  General Health State Questionnaire
EuroQoL 5 Dimensions | pre and post intervention and 6 and 12 months of follow up
  Health Related Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Principal Investigator — University of Malaga and Faculty of Health at the Queensland University of Technology
Locations (1):
- Patronato Municipal de Deportes de Torremolinos, Torremolinos, Málaga, Spain

REFERENCES:
- [Derived] Cuesta-Vargas AI, Gonzalez-Sanchez M. Changes in disability, physical/mental health states and quality of life during an 8-week multimodal physiotherapy programme in patients with chronic non-specific neck pain: a prospective cohort study. PLoS One. 2015 Feb 24;10(2):e0118395. doi: 10.1371/journal.pone.0118395. eCollection 2015. PMID 25710539